CLINICAL TRIAL: NCT02166918
Title: Multicenter Study on Factors Influencing Real-life Social Functioning of People With a Diagnosis of Schizophrenia
Brief Title: Factors Influencing Social Functioning of People With Schizophrenia
Acronym: PRIN2014
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: University of Turin, Italy (Other); University of Bari (Other); University of Genova (Other)
Responsible Party: Principal Investigator, Prof. Silvana Galderisi, Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 2010XP2XR4
Record Dates: First submitted 2014-03-19; First posted 2014-06-18 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Real-Life Functioning; Schizophrenia Endophenotypes
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — In all subjects a blood sample of 20 ml will be withdrawn from a peripheral vein for genetic analyses.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- patients with schizophrenia: 320 patients with a diagnosis of schizophrenia according to Diagnostic and Statistical Manual IV edition (DSM-IV) criteria, confirmed by the Structured Clinical Interview for DSM-IV - Patient Version (SCID -IP), will be included in the study.
- unaffected first-degree relatives: 240 unaffected first-degree relatives of the recruited patients (120 unaffected parents and 120 unaffected siblings)
- healthy control: 320 healthy control subjects.

SUMMARY:
In the last decades the impact of several variables on patients' social functioning has been investigated with conflicting findings. The involved variables might be grouped in three main categories: a) disease-related variables; b) personal resources; c) context-related factors. The present study is aimed to identify factors that affect most real-life functioning of subjects with schizophrenia and to assess negative and depressive symptoms, neurocognitive deficits and impairment of social cognition. Domains of negative symptoms and cognitive dysfunctions most associated with impairment of real-life functioning will be identified and appropriate data analyses will be carried out to define whether it has a direct or indirect impact on real-life functioning. The research units of Turin and Genua will also investigate the relationships between insight into the illness and real-life social functioning. The research unit of Genua will evaluate prevalence and course of depressive symptoms, insight impairment and neurocognitive deficits, and will define the relationships of these aspects with suicidal behavior and real-life social functioning. The Naples research unit n.1 will investigate the hypothesis that deficits of preattentive and perceptual functions underlie impaired social cognition and negative symptoms. An electrophysiological study will be carried out in which abnormalities of event-related components and gamma rhythm synchronization, relevant to preattentive and perceptual stages of information processing, will be studied as endophenotypes of the disorder.

The study will also investigate the heritability of disease-related variables by evaluating them in non-affected, first-degree relatives of subjects with schizophrenia. The research unit of Bari will test functionality of genetic variants relevant to dopaminergic signaling, that might confer risk for neurocognitive and related prefrontal dysfunction assessed by specific functional magnetic resonance imaging (fMRI) paradigms. The Naples research unit n. 6 will perform an association study between selected putative schizophrenia genes and specific psychometric, neurophysiological and neurocognitive schizophrenia endophenotypes; moreover, the research unit will search for de novo copy-number variations (CNV) as putative risk factors for schizophrenia or schizophrenia endophenotypes and for de novo protein-altering mutations that may contribute to the genetic component of schizophrenia endophenotypes. The Naples research unit n. 5 will be responsible for defining a standardized protocol for the assessment of medical comorbidities in subjects with schizophrenia. All psychiatric research units will contribute to assess the role of factors related to the context in modulating the impact of variables related to the disease on real-life social functioning.

DETAILED DESCRIPTION:
The study will last 36 months. The questionnaire for the assessment of physical health and medical conditions risk factors, as well as the manual concerning the procedures for screening and assessment of medical comorbidity, will be developed during the first three months of the study. The recruitment and assessment of all subjects will be completed within the first semester of the third year.

The analysis of data collected will be completed in the second semester of the third year.

PROCEDURES AND ASSESSMENT TOOLS In all subjects a blood sample of 20 ml will be withdrawn from a peripheral vein for genetic analyses.

1. Evaluation of aspects related to the disease. For all patients a clinical form will be filled in with data on age and type of disease onset, course of the disease and treatments. All available sources of information (patient, family, medical records and mental health workers) will be used to complete the form.

   The Premorbid Adjustment Scale (PAS) will be used to assess premorbid adjustment. It evaluates the achieved level of functioning before the onset of schizophrenia in four areas (social accessibility/isolation, peer relationships, ability to function outside the nuclear family, and capacity to form intimate social - sexual ties) during 4 periods of subject's life (childhood; early adolescence; late adolescence; adulthood), as well as the highest achieved global level of functioning. It comprises 26 items with a score ranging from 0 (healthiest end of the adjustment range) to 6 (indicating the least healthy end).

   General psychopathology and positive symptoms will be evaluated using the Positive and Negative Syndrome Scale (PANSS).

   Negative symptoms will be assessed using the Brief Negative Symptom Scale (BNSS). This scale includes 13 items and assesses 5 domains of negative symptoms: anhedonia, asociality, avolition, blunted affect and alogia, as well as a control item, not included in the negative domains, "Distress". For all items of the 5 domains higher scores are associated with greater impairment/presence of symptoms, while for the item Distress the highest score is associated with reduction or absence of negative emotions.

   Depressive symptoms will be investigated using the Calgary Depression Rating Scale (CDRS), a rating scale designed to assess the level of depression in people with schizophrenia. It includes 9 items (depression; hopelessness; self depreciation; guilty ideas of reference; pathological guilt; morning depression; early wakening; suicide; observed depression) with a score ranging from 0 (absent) to 3 (severe).

   The possible presence of extrapyramidal symptoms, whose assessment is required to exclude that the observed negative symptoms are secondary to them, will be verified by means of the St. Hans Rating Scale (SHRS), a multidimensional rating scale comprising four subscales: hyperkinesias, parkinsonism, akathisia and dystonia. Each subscale includes one or more items with a score ranging from 0 (absent) to 6 (severe).

   Neurocognitive functions will be evaluated by means of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB). The battery includes tests for the assessment of seven distinct cognitive domains: a) processing speed, b) attention/vigilance, c) working memory, d) verbal learning, e) visual learning, f) social cognition and g) reasoning and problem solving.

   The assessment of social cognition, partly included in the MCCB, will be completed using the Facial Emotion Identification Test and a theory of mind test The Awareness of Social Inference Test (TASIT). In the Facial Emotion Identification Test (FEIT), 55 faces are presented on a screen; the subject has to choose the facial emotion expressed by each face among 7 possibilities (anger, disgust, neutral, happiness, surprise, fear, sadness). The TASIT includes three sections: 1) Emotion Evaluation Test, that examines the ability to recognize basic emotions shown by other people, in which 28 vignettes are presented to the subject who has to choose the emotion expressed by a target actor from a multiple-choice array (surprise, happiness, anger, sadness, anxiety, disgust, neutral); 2) Test of Social Inference (Minimal), that evaluates the ability to perceive social inferences, specifically those involving the use of sarcasm; 15 vignettes are presented and the subject has to answer, for each vignette, four questions regarding, respectively, what one of the actors was "doing", what was he/she trying to "say", what was he/she "thinking" and what was he/she "feeling"; 3) Test of Social Inference (Enriched), that evaluates the ability to perceive social inferences involving lying and using sarcasm; 16 vignettes are presented and the same questions of the second section are asked.
2. Assessment of personal resources The evaluation of physical health status will be carried out through the application of a standardized protocol developed by the unit N. 5 of Naples.

The assessment of coping style will be made by means of the Coping Orientation to Problems Experienced inventory - Brief, including 28 items, divided into 14 scales: positive reframing, self-distraction, expression, use of instrumental support, active coping, denial, religion, humor, behavioral disengagement, use of emotional support, substance use, acceptance, planning, self-blame. The tool aims to capture a wide range of coping strategies in real life situations.

The evaluation of self-esteem will be carried out using the Self-Esteem Rating Scale (SERS), which assesses different aspects of the self-esteem, such as feeling socially and self-competent, being worth of respect, feeling intelligent and able to solve problems. SERS is composed of 40 items, with ratings on a 7-point Likert scale.

The recovery style will be evaluated using the Recovery Style Questionnaire. This self-administered instrument consists of 39 items that refer to the construct of continuity, ownership, responsibility, curiosity, education, help-seeking, blame, cause, optimism, impact, fear, liking and satisfaction. For each of them the person is categorized as sealer or integrator.

Resilience will be evaluated through the Resilience Scale for Adults (RSA). The RSA is a scale that provides a multidimensional assessment of resilience general characteristics. It includes 33 items that examine intra-and inter-personal protective factors thought to facilitate adaptation when facing psychosocial adversity. Factor analysis showed six factors: a) personal competence, b) positive perception of the future, c) social competence, d), personal structure, and) family cohesion, f) social resources.

The relationship with mental health services will be evaluated with the Service Engagement Scale (SES), which includes 16 items grouped into 4 subscales: a) availability, b) cooperation c) help seeking d) adherence to treatment. The person is given a score on a 4-point Likert scale. c) Evaluation of factors related to the context. For the evaluation of subject's family social - economic status the Social Economic Status will be used. The SES is based on: a) education and b) type of work. The educational level is measured on a 7-level scale (1=elementary school, 7=post-degree/specialization courses) and the type of work is rated on a 9-level scale (1=laborer, 9=high level managerial positions). To calculate the index the education level and the type of work of each parent is weighted.

The amount of social policies expenditure and the unemployment rate in the geographical macro-area (Northeast, Northwest, Central, South and Islands) will be taken from the latest Italian National Institute of Statistic (ISTAT) tables. The availability of a disability pension, and access to family and social incentives will be investigated through a social - demographic questionnaire developed ad hoc with which data on sex, age, marital status, schooling, housing, and luxuries habits will be also collected. For the evaluation of the social network the Social Network Questionnaire (SNQ) will be used. It is a self-administered questionnaire that evaluates the structural and qualitative aspects of the social network. It includes 15 items, grouped into 4 factors: a) quality and frequency of social contacts; b) practical social support; c) emotional support, d) quality of an intimate relationship. Each item is rated on a scale from 1 "never" to 4 "always". The evaluation of the stigma associated with mental illness will be carried out using two instruments: the Internalized Stigma of Mental Illness (ISMI), which will be administered to all patients and evaluates the experience of stigma and internalized self-rejection, and the Perceived Devaluation and Discrimination Scale (PDD), which measures the perceived stigma, i.e., the attitudes of the general population with respect to mental disorders, which will be administered to all subjects. The ISMI is a scale that includes 29 items and 5 subscales for self-assessment of subjective experience of stigma. Each item is rated on a 4-level Likert scale, where higher scores indicate greater levels of internalized stigma. The PDD includes 12 items, each of whom is rated on a 5-level Likert scale, with higher scores indicating greater stigma.

d) Assessment of functional capacity and real-life functioning The functional capacity will be evaluated using the short version of the Performance-based Skills Assessment, University of California, San Diego (UCSD) , a performance-based instrument that investigates two areas: Financial Skills (counting money, counting change and paying bills) and Communication Skills (to dial a telephone number for emergency, for information, dial a telephone number from memory; to reschedule an appointment by telephone; to understand and to remember the instructions on a Medical Doctor Appointment Letter). Individual real-life functioning will be assessed by the Specific Level of Function Scale (SLOF), a hybrid instrument that explores many aspects of functioning and is based on judgments by a caregiver/operator (or the direct observation) of behavior and functioning of patients. It consists of 43 items and includes the following domains: a) physical efficiency; b) skills in self-care; c) interpersonal relationships; d) social acceptability; e) community activities (e.g., shopping, using public transportation); f) working abilities. The scale that assesses "Personal and Social Functioning" (PSF) will be also used; it evaluates the areas of self-care, socially useful activities, personal and social relationships and disturbing and aggressive behaviors.

GENETIC ASSOCIATION ANALYSES WITH THE PHENOTYPES OF INTEREST The Naples research unit n. 6 will perform an association study between selected putative schizophrenia genes and specific psychometric, neurophysiological and neurocognitive schizophrenia endophenotypes; moreover, the research unit will search for de novo copy-number variations (CNV) as putative risk factors for schizophrenia or schizophrenia endophenotypes and for de novo protein-altering mutations that may contribute to the genetic component of schizophrenia endophenotypes.

STATISTICAL ANALYSIS OF DATA To identify the factors that affect most real-life functioning of people diagnosed with schizophrenia multiple regression statistical models will be used. Real-life functioning and functional capacity indices will be defined as dependent variables. The three blocks of variables, i.e. disease-related variable, personal resources and context-related variables, will be the independent variables or predictors. structural equation model (SEM), that according to some authors is robust against the problem of multicollinearity occurring in a regression model when there is a linear correlation among the independent variables, will be used. This analysis allows to draw assumptions on the causality between the variables and, based on path analysis o identify potential factors mediating and moderating the relationships between dependent and independent variables. The explored models will be subsequently tested with confirmatory analyses.

Estimated sample size for this analysis is of at least 5 independent observations for each index in the model. Therefore, by including in the model: 3 demographic indices (age, sex and education), 15 variables related to the disease (PANSS-general and PANSS-positive subscale scores, 2 negative symptom domains derived from BNSS, 6 cognitive domains from the MCCB, 4 indices of social cognition, derived from the specific section of the MCCB, TASIT and FEIT, the total score for depression on the Calgary scale), 36 indices related to the personal resources (6 factors of Resilience, 14 Coping factors, 13 Recovery styles factors, 1 score for Self-Esteem, 1 index of relationship with mental health services, 1 physical health index) and 10 related to the context (1 index of economic status, 5 indices of financial opportunities and work/family and social incentives, 2 stigma indices, 2 social network factors), for a total of 64 indices, it is estimated that an appropriate sample of patients will be 64x5=320 subjects.

The effects of dichotomous variables (eg, gender) and ordinal (eg, social class) will be assessed with one- or multiple-way analyses of variance. The analyses will be conducted using the Statistical Package for Social Science (SPSS).

ELIGIBILITY:
Inclusion Criteria for patients recruited from those attending the outpatient units of the University Psychiatric Clinics of Naples, Turin, Genova and Bari:

1. diagnosis of schizophrenia according to DSM-IV, confirmed with the Structured Clinical Interview for DSMIV - Patient version (SCID-I-P),
2. age between 18 and 65 years

Exclusion Criteria for patients:

1. a history of head trauma with loss of consciousness,
2. neurological disease,
3. history of alcoholism or substance abuse in the last six months,
4. pregnancy,
5. inability to provide informed consent,
6. moderate or severe mental retardation,
7. changes in antipsychotic therapy and hospitalization for exacerbation of symptoms in the 3 months prior to inclusion in the study.

Exclusion criteria for unaffected relatives and healthy controls:

1. a positive personal history of psychiatric disorders and/or
2. a family history of mood or psychotic disorders or hospitalization in a psychiatric hospital.
3. any degree of mental retardation
4. current use of medications with central nervous system effects.
5. those listed in a-e for patients

The Structured Clinical Interview for DSM IV Non Patients Version (SCID-NP-I) and the SCID II will be administered to both healthy controls and family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three-hundred-twenty patients (80 in each of the 4 recruitment units) with a diagnosis of schizophrenia according to DSM-IV criteria, confirmed by the Structured Clinical Interview for DSM-IV - Patient Version (SCID -IP), will be included in the study. One-hundred-twenty unaffected parents of the recruited patients (15 pairs of parents in each center), 120 unaffected siblings and 320 healthy control subjects, meeting the criteria listed below, will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Factors contributing to real life impairment in schizophrenia | 36 months
  The primary objective of this study is to identify factors that affect most real-life functioning of patients with schizophrenia and define their relative contribution. To these aims, disease-related variables, personal resources and context-related factors will be evaluated as independent variables, while real-life functioning of the examined subjects will be the dependent variable. For each factor we will define whether its impact on real-life functioning is direct or indirect, i.e. mediated by the effects on another factor, in its turn associated with functioning.

SECONDARY OUTCOMES:
Relation between impairment of social cognition, negative symptoms and preattentive and perceptual deficits | 36 months
  Verify, in a subgroup of subjects, the hypothesis that the impairment of some aspects of social cognition and negative symptoms, in particular the factor "anhedonia/asociality/avolition", are related to preattentive and perceptual deficits. Verify, in a subgroup of subjects, the impact of poor insight on social functioning of patients.
Associations between schizophrenia candidate genes and endophenotypes of the disorder | 36 months
  Demonstrate, in a subgroup of subjects, the existence of associations between schizophrenia candidate genes and endophenotypes of the disorder, in particular: associations between functional genetic variants related to dopaminergic transmission and indices of neurocognitive and prefrontal dysfunction, evaluated by functional MRI during a working memory task and associations between polymorphisms of genes regulating dopaminergic and glutamatergic transmission and electrophysiological endophenotypes
Prevalence of physical comorbidities | 36 months
  Prevalence of physical comorbidities in individuals with schizophrenia using a standardized protocol developed for this purpose
Severity of physical comorbidities | 36 months
  Investigate the severity of physical comorbidities in individuals with schizophrenia using a standardized protocol developed for this purpose

OTHER OUTCOMES:
Prevalence of depressive symptoms in individuals with schizophrenia | 36 months
  Investigate, in a subgroup of subjects, the prevalence of depressive symptoms and the influence of these aspects on the emergence of suicidal behaviors.
Course of depressive symptoms in individuals with schizophrenia | 36 months
  Investigate, in a subgroup of subjects, the course of depressive symptoms and the influence of these aspects on the emergence of suicidal behaviors.
Prevalence of poor insight and neurocognitive deficits in individuals with schizophrenia | 36 months
  Investigate, in a subgroup of subjects, the prevalence poor insight and neurocognitive deficits, and the influence of these aspects on real life functioning
Course of poor insight and neurocognitive deficits in individuals with schizophrenia | 36 months
  Investigate, in a subgroup of subjects, the course poor insight and neurocognitive deficits, and the influence of these aspects on real life functioning

CONTACTS AND LOCATIONS:
Overall Officials: Mario Maj, MD, PhD, Study Director — University of Naples, SUN
Locations (4):
- Italy (4):
  - Psychiatric University Hospital, University of Naples, SUN, Napoli, Napoli
  - University of Bari ITALY, Bari
  - University of Genova ITALY, Genova
  - University of Torino ITALY, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monteleone P, Bifulco M, Di Filippo C, Gazzerro P, Canestrelli B, Monteleone F, Proto MC, Di Genio M, Grimaldi C, Maj M. Association of CNR1 and FAAH endocannabinoid gene polymorphisms with anorexia nervosa and bulimia nervosa: evidence for synergistic effects. Genes Brain Behav. 2009 Oct;8(7):728-32. doi: 10.1111/j.1601-183X.2009.00518.x. Epub 2009 Jun 26. PMID 19659925
- [Background] Galderisi S, Bucci P, Mucci A, Kirkpatrick B, Pini S, Rossi A, Vita A, Maj M. Categorical and dimensional approaches to negative symptoms of schizophrenia: focus on long-term stability and functional outcome. Schizophr Res. 2013 Jun;147(1):157-162. doi: 10.1016/j.schres.2013.03.020. Epub 2013 Apr 19. PMID 23608244
- [Background] Maj M. Understanding the pathophysiology of schizophrenia: are we on the wrong or on the right track? Schizophr Res. 2011 Apr;127(1-3):20-1. doi: 10.1016/j.schres.2011.01.002. Epub 2011 Feb 1. No abstract available. PMID 21277744
- [Background] Maj M. The rights of people with mental disorders: WPA perspective. Lancet. 2011 Oct 29;378(9802):1534-5. doi: 10.1016/S0140-6736(11)60745-9. Epub 2011 Oct 16. No abstract available. PMID 22008423
- [Background] Monteleone P, Martiadis V, Maj M. Management of schizophrenia with obesity, metabolic, and endocrinological disorders. Psychiatr Clin North Am. 2009 Dec;32(4):775-94. doi: 10.1016/j.psc.2009.08.003. PMID 19944883
- [Background] Maj M. Physical health care in persons with severe mental illness: a public health and ethical priority. World Psychiatry. 2009 Feb;8(1):1-2. doi: 10.1002/j.2051-5545.2009.tb00196.x. No abstract available. PMID 19293947
- [Background] Galderisi S, Maj M. Deficit schizophrenia: an overview of clinical, biological and treatment aspects. Eur Psychiatry. 2009 Dec;24(8):493-500. doi: 10.1016/j.eurpsy.2009.03.001. Epub 2009 Jun 23. PMID 19553087
- [Background] Galderisi S, Davidson M, Kahn RS, Mucci A, Boter H, Gheorghe MD, Rybakowski JK, Libiger J, Dollfus S, Lopez-Ibor JJ, Peuskens J, Hranov LG, Fleischhacker WW; EUFEST group. Correlates of cognitive impairment in first episode schizophrenia: the EUFEST study. Schizophr Res. 2009 Dec;115(2-3):104-14. doi: 10.1016/j.schres.2009.09.022. Epub 2009 Oct 12. PMID 19822407